CLINICAL TRIAL: NCT01429506
Title: Effect of Laparoscopic Sleeve Gastrectomy and Intensive Medical Management in Obese Type 2 Diabetes
Brief Title: Efficacy of Laparoscopic Sleeve Gastrectomy and Intensive Medical Management in Obese Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, Professor, Department of endocrinology, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 922861
Record Dates: First submitted 2011-09-04; First posted 2011-09-07 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus; Obesity
Keywords: Sleeve gastrectomy; Intensive medical management
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleeve gastrectomy (Active Comparator): Will undergo laparoscopic sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy
- Intensive medical management (Active Comparator): Will receive VLCD, exenatide, metformin, insulin detemir
  Interventions: Drug: Intensive medical management

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Sleeve gastrectomy
  Other Names: Bariatric surgery; Laparoscopic sleeve gastrectomy
  Arms: Sleeve gastrectomy
Drug: Intensive medical management — Exenatide 10 mcg BD, Metformin 2-3 gm/day, 800 Kcal diet
  Arms: Intensive medical management

SUMMARY:
In this the investigators will be comparing the effects of Laparoscopic sleeve gastrectomy with intensive medical management on weight and metabolic parameters.

DETAILED DESCRIPTION:
Intensive medical management will include

1. VLCD
2. Physical activity
3. Exenatide
4. Metformin
5. Insulin detemir

ELIGIBILITY:
Inclusion Criteria:

Type 2 Diabetics with

1. BMI ≥ 27.5 kg/m2
2. HbA1c 7-10%
3. Age 20-70 years

Exclusion Criteria:

1. Prior gastric surgery
2. Pregnancy and lactation
3. renal disease (GFR < 60 ml/min)
4. Pancreatitis
5. Symptomatic gallstone disease
6. Active malignancy
7. Secondary causes of obesity ( Cushing's syndrome, uncontrolled Hypothyroidism)
8. Severe psychiatric illness
9. Allergic reaction to exenatide

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
weight loss | 6 months
  weight loss at 6 months after the start of intervention

SECONDARY OUTCOMES:
glycemic control | 6 months
  HbA1c and glucose profile

CONTACTS AND LOCATIONS:
Overall Officials: Anil Bhansali, DM, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India